CLINICAL TRIAL: NCT05784402
Title: A Randomised Study to Investigate Steady State Semaglutide Exposure of a New Formulation of Oral Semaglutide in Healthy Participants
Brief Title: A Research Study to Compare How Much Semaglutide is Found in the Blood With Different Tablets of Oral Semaglutide in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4891; U1111-1279-6289 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sequence A: Semaglutide J-Semaglutide C-Semaglutide J (Experimental): After 6 weeks of run-in dose escalation period participants will orally receive semaglutide J at dose level 1 once daily for 4 weeks followed by semaglutide C once daily for next 4 weeks and thereafter semaglutide J at dose level 3 once daily for next 4 weeks.
  Interventions: Drug: Semaglutide J; Drug: Semaglutide C
- Sequence B: Semaglutide C-Semaglutide J-Semaglutide J (Experimental): After 6 weeks of run-in dose escalation period participants will orally receive semaglutide C once daily for 4 weeks followed by semaglutide J at dose level 2 once daily for next 4 weeks and thereafter semaglutide J at dose level 4 once daily for next 4 weeks.
  Interventions: Drug: Semaglutide J; Drug: Semaglutide C
- Sequence C: Semglutide J-Semaglutide J-Semaglutide C (Experimental): After 6 weeks of run-in dose escalation period participants will orally receive semaglutide J at dose level 1 once daily for 4 weeks followed by semaglutide J at dose level 3 once daily for next 4 weeks and thereafter semaglutide C (2x dose) once daily for next 4 weeks.
  Interventions: Drug: Semaglutide J; Drug: Semaglutide C
- Sequence D: Semaglutide J-Semaglutide C-Semaglutide J (Experimental): After 6 weeks of run-in dose escalation period participants will orally receive semaglutide J at dose level 2 once daily for 4 weeks followed by semaglutide C (2x dose) once daily for next 4 weeks and thereafter semaglutide J at dose level 4 once daily for next 4 weeks.
  Interventions: Drug: Semaglutide J; Drug: Semaglutide C

INTERVENTIONS:
Drug: Semaglutide J — Participants will receive oral semglutide J at dose level 1 and 3 in treatment sequence A and C; and at dose level 2 and 4 in treatment sequence B and D.
Drug: Semaglutide C — Participants will receive oral semglutide C in treatment sequence A and B; and at semglutide C at 2x dose level in treatment sequence C and D.

SUMMARY:
In this study, a known investigational medicine called 'semaglutide' will be tested in 2 different tablet versions. In addition to semaglutide, the tablet versions contain different helping agents in different amounts. Both tablet versions have a helping agent called SNAC. The main aim of this study is to investigate semaglutide of 4 different doses in a new tablet by determining the amount of semaglutide in the blood and compare the concentration in the blood for the new tablet with the tablet currently investigated in a phase 3b study (current version). For this purpose, the amount of semaglutide in the blood will be measured after multiple doses of semaglutide, at different doses. Which doses participant will get will be decided by chance. The study will have 4 groups (A-D) and will include up to 260 participants. The doses participant get depends on the group they are (enrolled) in. All four groups will be receiving the investigational medicine for 15 weeks in total. Group A will start testing the dose level 1 (new tablet) for 5 weeks. Then receiving the current tablet of semaglutide C for 5 weeks and then testing the dose level 3 (new tablet) for 5 weeks. Group B will start receiving the current tablet semaglutide C for 5 weeks and then testing the dose level 2 (new tablet) in 5 weeks and dose level 4 (new tablet) in 5 weeks. Group C will start testing the dose level 1 (new tablet) and dose level 3 (new tablet) for 5 weeks each and then receiving the current tablet of semaglutide C (2x dose) for 5 weeks. Group D will start testing the dose level 2 (new tablet) for 5 weeks. Then receiving the current tablet of semaglutide C (2x dose) for 5 weeks and then testing the dose level 4 (new tablet) for 5 weeks. Participants will be receiving doses of semaglutide for 6 weeks before being assigned to one of the 4 groups (A-D) to reduce the risk of side effects. Participants cannot choose which group they want to be in, and they can only participate in one group in this study. Participant will get one tablet to be taken by mouth each day for approximately 21 weeks. The tablet should be taken in the morning together with no more than half a glass of water (120 milliliter [mL]), after an overnight fast of at least 6 hours (no food or drinks). Water is also not allowed from 2 hours before dosing. After dosing, participant must begin breakfast no earlier than 30 minutes and no later than 35 minutes after having taken tablet. The study will last for about 30 weeks in total for each participant. This includes a screening period (up to 4 weeks), a dose escalation period (6 weeks), an investigational treatment period (15 weeks) and a follow-up period (5 weeks after last dose). The planned duration a participant can receive trial product is 21 weeks. Participant should not take any prescription or non-prescription medicines (including herbal products) within 14 days prior to the screening visit (visit 1) and until the follow-up visit, except for birth control, routine vitamins, medicines applied on the skin, and occasional use of acetaminophen or ibuprofen (a mild pain killer). No oral medication (medicine taken by mouth) can be taken from 2 hours before and until 30 minutes after each dosing with semaglutide. Women cannot take part if pregnant, breast-feeding or planning to become pregnant during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 23.0 and 34.9 kilograms per meter square (kg/m^2) (both inclusive) at screening
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using highly effective contraceptive method
* Any disorder, which in the investigator's opinion might jeopardise participant's safety or compliance with the protocol
* Use of prescription medicinal products or non-prescription drugs, except highly effective contraceptives, routine vitamins, topical medication not reaching the systemic circulation and occasional use of paracetamol (acetaminophen) and ibuprofen within 14 days before screening
* Presence of clinically significant gastrointestinal disorders potentially affecting absorption of drugs, as judged by the investigator

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 264 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
AUC0-24h,semaglutide,SS; area under the semaglutide plasma concentration-time curve during a dosing interval at steady state | From 0 to 24 hours after dosing on days 77, 112 and 147
  Measured in hours*nanomoles per liter (h*nmol/L).

SECONDARY OUTCOMES:
Cmax,0-24h.semaglutide,SS; maximum observed plasma concentration of semaglutide at steady state | From 0 to 24 hours after dosing on days 77, 112 and 147
  Measured in nanomoles per liter (nmol/L).
tmax,0-24h,semaglutide,SS; Time to maximum semaglutide plasma concentration at steady state | From 0 to 24 hours after dosing on days 77, 112 and 147
  Measured in hours (h).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (3):
- United States (2):
  - Altasciences Clinical LA, Inc., Cypress, California
  - Altasciences Clinical Kansas, Inc., Kansas City, Kansas
- Altasciences Clinical Company, Inc, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com